CLINICAL TRIAL: NCT01565655
Title: A Phase 2b, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Dose-Finding, Multi-Center Study to Evaluate the Safety and Efficacy of ASP015K in Moderate to Severe Rheumatoid Arthritis Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of ASP015K in Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 015K-CL-RA22; 2011-006020-20 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; ASP015K
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ASP015K lowest dose (Experimental): ASP015K lowest dose once daily
  Interventions: Drug: peficitinib
- ASP015K low dose (Experimental): ASP015K low dose once daily
  Interventions: Drug: peficitinib
- ASP015K medium dose (Experimental): ASP015K medium dose once daily
  Interventions: Drug: peficitinib
- ASP015K high dose (Experimental): ASP015K high dose once daily
  Interventions: Drug: peficitinib
- Placebo (Placebo Comparator): Matching placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K
  Arms: ASP015K high dose; ASP015K low dose; ASP015K lowest dose; ASP015K medium dose
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ASP015K in moderate to severe rheumatoid arthritis (RA) subjects

DETAILED DESCRIPTION:
Subjects will take ASP015K or matching placebo orally with food for 12 weeks after randomization. Potential subjects who have previously used disease-modifying antirheumatic drugs (DMARDs) and/or biologic agents may be eligible to participate after completing a washout period. Subjects who complete the 12-week dosing period in this study may be eligible to participate in a long-term, open-label Extension Study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 tender/painful joints; ≥ 6 swollen joints
* C-Reactive Protein (CRP) of ≥ 0.8 mg/dL or Erythrocyte Sedimentation Rate (ESR) of ≥ 28 mm/hr
* Subject meets the ACR 1991 Revised Criteria for Global Functional Status in RA Class I, II or III at Screening and Baseline
* Use of non-steroidal anti-inflammatory drugs [NSAIDs], cyclooxygenase-2 (COX-2) inhibitors, or oral corticosteroids for the treatment of RA must be stable for at least 28 days prior to start of the study
* Male and female subjects must be willing to comply with contraception requirements as well as restrictions regarding egg and sperm donation
* Female subject must not be breastfeeding at Screening or during the study period, and for 60 days after the final study drug administration
* Subject agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

* Positive Mycobacterium tuberculosis (TB) test within 90 days of Screening
* Abnormal chest x-ray indicative of an acute or chronic infectious process or malignancy
* Receipt of live or live attenuated virus vaccination within 30 days prior to the first dose of study drug
* Known history of positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody or history of a positive test for human immunodeficiency virus (HIV) infection
* History of any other autoimmune rheumatic disease, other than Sjogren's syndrome
* Previous history of clinically significant infections or illness (requiring hospitalization or requiring parenteral therapy) within 90 days of the Baseline visit, or a history of any illness that would preclude participation in the study
* History of any malignancy, except for successfully treated basal or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix.
* Does not meet specified washout criteria for the following RA medications: gold, azathioprine, minocycline, penicillamine, etanercept, certolizumab, adalimumab, golimumab, infliximab, cyclophosphamide, and leflunomide
* Previous intolerance to Janus kinase (JAK) inhibitors
* Receipt of intra-articular or parenteral corticosteroid within 28 days prior to the first dose of study drug or is currently taking > 30 mg oral morphine (or narcotic equivalent) per day
* Receipt of plasma exchange therapy within 60 days prior to the start of study drug
* Receipt of any investigational agent within 30 days or 5 half-lives, whichever is longer, prior to first dose of study drug
* Receipt of medications that are CYP3A substrates with narrow therapeutic range within 14 days prior to first dose of study drug
* History of heart failure, defined as New York Heart Association (NYHA) grade 3 or greater
* History of long QT syndrome or prolonged QT interval
* Any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, or infectious disease, or any ongoing illness which would make the subject unsuitable for the study
* Subject has any condition possibly affecting oral absorption (e.g., gastrectomy, other malabsorption syndromes, or clinically significant diabetic gastroenteropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving American College of Rheumatology Criteria 20 (ACR 20) response | Week 12
Trough plasma concentration of ASP015K and metabolite(s) | up to Week 12 (6 time points)

SECONDARY OUTCOMES:
Percentage of subjects achieving ACR 50 response | Week 12
Percentage of subjects achieving ACR 70 response | Week 12
Change from baseline in Disease Activity Score using 28 joint count and C Reactive Protein (DAS28-CRP) | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (38):
- United States (19):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Stanford University School of Medicine, Palo Alto, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Arthritis Associates of Colorado Springs, Colorado Springs, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Arthritis Associates, Orlando, Florida
  - Illinois Bone & Joint Institute; LLC, Morton Grove, Illinois
  - Deerbrook Medical Asssociates, Vernon Hills, Illinois
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - PMG Research, Hickory, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clincal Research Center of Reading, Wyomissing, Pennsylvania
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Austin Rheumatology Research PA, Austin, Texas
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Bulgaria (3):
  - MHAT Burgas, Burgas
  - MHAT Plovdiv AD, Plovdiv
  - MHAT "Sv. Ivan Rilski", Sofia
- Czechia (4):
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Praha-Nusle
  - MEDICAL PLUS, s.r.o. or REVMACENTRUM UH, s.r.o., Uherské Hradiště
  - PV-MEDICAL s.r.o., Zlín
- Hungary (5):
  - Rethy Pal Korhaz es Rendelointezet, Békéscsaba
  - Budai Irgalmasrendi Korhaz, Budapest
  - Orszgos Reumatolgiai s Fizioterpis Intzet, Budapest
  - Revita Clinic Rheumatology, Budapest
  - Kenezy Hospital Institute of Clinical Pharmacology, Debrecen
- Mexico (3):
  - Cliditer S.A. de C.V., Mexico City, Mexico City
  - Dr Javier Orozco Alcala Private Doctor´s office, Guadalajara
  - Centro de Investigacion Clinica de Morelia, S.C., Morelia
- Poland (4):
  - Szpital Uniwersytecki nr. 2 im. Dr. Jana Biziela, Bydgoszcz
  - NZOZ Centrum Medyczne ProMiMed, Krakow
  - Zespol Poradni Specjalistycznych, REUMED sp. Zo.o, Lublin
  - ARS Rheumatica, Warsaw

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028
- [Derived] Genovese MC, Greenwald M, Codding C, Zubrzycka-Sienkiewicz A, Kivitz AJ, Wang A, Shay K, Wang X, Garg JP, Cardiel MH. Peficitinib, a JAK Inhibitor, in Combination With Limited Conventional Synthetic Disease-Modifying Antirheumatic Drugs in the Treatment of Moderate-to-Severe Rheumatoid Arthritis. Arthritis Rheumatol. 2017 May;69(5):932-942. doi: 10.1002/art.40054. PMID 28118538
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=323